CLINICAL TRIAL: NCT05535803
Title: Treatment of Laryngotracheal Stenosis Using Autologous Olfactory-mucosa-derived Mesenchymal Stem Cells
Brief Title: Treatment of Laryngotracheal Stenosis Using Mesenchymal Stem Cells
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: The Republican Center for Research and Practice in Otolaryngology (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_MSCStenosis
Record Dates: First submitted 2022-08-26; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Tracheal Stenosis; Laryngeal Stenosis
Keywords: mesenchymal stem cells; Tracheal/Laryngeal Stenosis
MeSH Terms: conditions — Tracheal Stenosis; Laryngostenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with tracheal/laryngeal stenosis receiving standard treatment and stem cells (Experimental): Patients with tracheal/laryngeal stenosis receiving standard surgical treatment and mesenchymal stem cells
  Interventions: Biological: Olfactory mucosa-derived mesenchymal stem cells; Other: Patients treated according to current clinical protocols
- Patients with tracheal/laryngeal stenosis receiving standard treatment (Active Comparator): Patients with tracheal/laryngeal stenosis receiving standard surgical treatment
  Interventions: Other: Patients treated according to current clinical protocols

INTERVENTIONS:
Biological: Olfactory mucosa-derived mesenchymal stem cells — Autologous olfactory mucosa-derived mesenchymal stem cells
  Arms: Patients with tracheal/laryngeal stenosis receiving standard treatment and stem cells
Other: Patients treated according to current clinical protocols — Patients treated according to current clinical protocols

SUMMARY:
The trial evaluates the safety and efficacy of the olfactory mucosa-derived mesenchymal stem cells based therapy for the patients with chronic laryngeal and tracheal stenosis

DETAILED DESCRIPTION:
Trial evaluating the safety and efficacy of olfactory mucosa-derived mesenchymal stem cells based therapy for the patients with chronic laryngeal and tracheal stenosis with/without cartilage defects

Mesenchymal stem cells are obtained from tissue biopsy of olfactory mucosa using explant method. Biomass of autologous mesenchymal stem cells in 10% human albumin solution is injected submucosally around and over the tissue after removal of a granuloma tissue during surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

-confirmed diagnosis of chronic laryngeal or tracheal stenosis;

Exclusion Criteria:

* refuse of patient to participate in the trial;
* acute infectious diseases;
* chronic mental disorders with severe manifestations;
* pregnancy/lactation;
* intercurrent severe chronic diseases;
* HIV, Hepatites B/C;
* active tuberculosis;
* alcohol use disorder/drug addiction;
* cachexia of any origin;
* malignant neoplasms.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients who didn't require the repeated surgical interventions | 1 year
  Relative number of patients who didn't require the repeated surgical interventions after MSC therapy

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Hancharou, Dr, Study Director — Institute for biophysics and cellular engineering NAS of Belarus; Elvira Strinkevich, Dr, Study Director — The Republican Center for Research and Practice in Otolaryngology; Valery Chekan, Dr, Study Director — The Republican Center for Research and Practice in Otolaryngology
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No